CLINICAL TRIAL: NCT02529254
Title: Video Coaching as an Efficient Teaching Method for Surgical Residents A Randomized Control Trial
Brief Title: Video Coaching as an Efficient Teaching Method for Surgical Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Pierre Dubé, Assistant director of clinical research, Chief of general surgery, Program director of general surgery., Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Surgery video coaching 15006
Record Dates: First submitted 2015-07-29; First posted 2015-08-20 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: post graduate surgical education; video coaching; Surgical education; coaching

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video coaching (Experimental): 14 residents in general surgery from PGY-1(post graduate year-1) to PGY-4 Block randomized to the intervention group who will receive a 30 minute video coaching session as the intervention
  Interventions: Behavioral: Video coaching session
- Control (No Intervention): 14 residents in general surgery from PGY-1 to PGY-4 block randomized to the control group

INTERVENTIONS:
Behavioral: Video coaching session — A 30 minute video coaching session with a surgeon in witch the residaent and coach visualise the filmed anastomosis and where the surgeon gives constructive feedback.
  Arms: Video coaching

SUMMARY:
The purpose of this study is to determine if video coaching is an efficient way of teaching surgical skills outside of the operating room for surgical residents.

DETAILED DESCRIPTION:
Coaching relates to a cooperative process between a coach and a coachee, which includes "providing objective and constructive feedback to help a [coachee] recognize what works and what can be improved.

In our study the investigators will be filming general surgery residents while making a side to side anastomosis on a dog's cadaveric small bowel. Half of the participants will be randomized in the intervention group and will take part in a half hour coaching session with a surgeon. In this coaching session both resident and surgeon will watch the resident's filmed anastomosis and constructive feedback will be given by the surgeon. An inanimate model of bowel anastomosis will be available at the moment of the coaching to allow the surgeon to demonstrate the desired improvements.

Once all the residents in the intervention group will have completed their coaching session, both control and intervention group will be filmed making a second side to side anastomosis.

All the video taken will then be pooled in a random order. A blinded surgeon will then analyse each video taken with the objective structured assessment of technical skills (OSATS) tool.

The hypothesis is that the residents who received an half-hour coaching session will have significantly improved their OSATS score compared to the control group between the first and second anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Residents from PGY-1 to PGY-4 in general surgery at Université de Montreal

Exclusion Criteria:

* PGY-5 in general surgery at université de Montreal ( because they are studying for their Board exams )
* Did no sing consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in (Objective structured assessment of technical skills) OSATS score at baseline and after the coaching session. | assessed at both first and second filmed anastomosis for both groups with about 1 month apart.

SECONDARY OUTCOMES:
Resident satisfaction questionnaire | Once every resident has completed his coaching session about two weeks after the first anastomosis.
  Questionnaire aiming to know if video coaching is something the participants think is useful.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael L Soucisse, MD, Principal Investigator
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Background] Singh P, Aggarwal R, Tahir M, Pucher PH, Darzi A. A randomized controlled study to evaluate the role of video-based coaching in training laparoscopic skills. Ann Surg. 2015 May;261(5):862-9. doi: 10.1097/SLA.0000000000000857. PMID 25185469
- [Background] Martin JA, Regehr G, Reznick R, MacRae H, Murnaghan J, Hutchison C, Brown M. Objective structured assessment of technical skill (OSATS) for surgical residents. Br J Surg. 1997 Feb;84(2):273-8. doi: 10.1046/j.1365-2168.1997.02502.x. PMID 9052454
- [Background] Greenberg CC, Ghousseini HN, Pavuluri Quamme SR, Beasley HL, Wiegmann DA. Surgical coaching for individual performance improvement. Ann Surg. 2015 Jan;261(1):32-4. doi: 10.1097/SLA.0000000000000776. No abstract available. PMID 24887977
- [Background] Bonrath EM, Dedy NJ, Gordon LE, Grantcharov TP. Comprehensive Surgical Coaching Enhances Surgical Skill in the Operating Room: A Randomized Controlled Trial. Ann Surg. 2015 Aug;262(2):205-12. doi: 10.1097/SLA.0000000000001214. PMID 25822691